CLINICAL TRIAL: NCT04193202
Title: A Phase 3b Randomized, Double-blind, Placebo Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Gefapixant in Adult Participants With Recent Onset Chronic Cough
Brief Title: Efficacy and Safety of Gefapixant (MK-7264) in Adult Participants With Recent Onset Chronic Cough (MK-7264-043)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7264-043; MK-7264-043 (Other: Merck Protocol Number); 2019-002308-42 (EudraCT Number)
Record Dates: First submitted 2019-12-09; First posted 2019-12-10 (Actual); Results first posted 2022-10-14 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Chronic Cough
Keywords: Cough; Respiration disorders; Respiratory tract diseases; Signs and symptoms, respiratory; Signs and symptoms
MeSH Terms: conditions — Chronic Cough; Cough; Respiration Disorders; Respiratory Tract Diseases; Signs and Symptoms, Respiratory; Signs and Symptoms | interventions — Gefapixant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gefapixant (Experimental): Participants will receive gefapixant at a dose of 45 mg administered as an oral tablet twice daily for 12 weeks.
  Interventions: Drug: Gefapixant
- Placebo (Placebo Comparator): Participants will receive placebo matching gefapixant, administered as an oral tablet twice daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gefapixant — Administered twice daily as an oral tablet of 45 mg
  Other Names: MK-7264
  Arms: Gefapixant
Drug: Placebo — Administered twice daily as a placebo oral tablet matching gefapixant
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of gefapixant in participants with recent onset chronic cough (duration >8 weeks after onset of cough symptoms) for <12 months and a diagnosis of refractory or unexplained chronic cough. The primary hypothesis is that gefapixant is superior to placebo in improving cough-related quality of life measured as change from baseline in the Leicester Cough Questionnaire (LCQ) total score at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Chest radiograph or CT thorax (within 1 year of Screening/Visit 1 and after the onset of chronic cough) not demonstrating any abnormality considered to be significantly contributing to the chronic cough or any other clinically significant lung disease, in the opinion of the principal investigator or the subinvestigator
* Has chronic cough (defined as duration of >8 weeks after onset of cough symptoms) for <12 months prior to the screening visit (<14 months after onset of cough symptoms)
* Has a diagnosis of refractory chronic cough or unexplained chronic cough
* Female participants are not pregnant, not breastfeeding, not of childbearing potential, or agree to follow contraceptive guidance

Exclusion Criteria:

* Is a current smoker
* Has given up smoking within 12 months of screening
* Is a former smoker with a smoking history greater than 20 pack-years (1 pack of 20 cigarettes per day for 20 years)
* Has a history of respiratory tract infection or recent change in pulmonary status within 4 weeks of screening
* Has a history of chronic bronchitis, defined as cough that produces >1 tablespoon of phlegm, that occurs every day for at least 3 months in a row
* Has a history of malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or cervical cancer
* Is a user of recreational or illicit drugs or a recent history (within the last year) of drug or alcohol abuse
* Has a history of anaphylaxis or cutaneous adverse drug reaction to sulfonamide-containing drugs
* Has a known allergy to gefapixant or its excipients
* Has donated or lost ≥1 unit (~300 mL) of blood within 8 weeks prior to first dose of gefapixant
* Has previously received gefapixant
* Is currently participating or has participated in an interventional clinical study within 30 days of participating in this current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (91):
- United States (15):
  - Pulmonary Associates, PA ( Site 0016), Phoenix, Arizona
  - Center for Clinical Trials, LLC ( Site 0035), Paramount, California
  - Springfield Clinic, LLP ( Site 0018), Springfield, Illinois
  - Chesapeake Clinical Research, Inc ( Site 0037), White Marsh, Maryland
  - Albuquerque Clinical Trials ( Site 0030), Albuquerque, New Mexico
  - Montefiore Einstein Center ( Site 0022), The Bronx, New York
  - American Health Research ( Site 0047), Charlotte, North Carolina
  - Clinical Research Institute of Southern Oregon, PC ( Site 0028), Medford, Oregon
  - Northwest Research Center ( Site 0039), Portland, Oregon
  - AAPRI Clinical Research Institute ( Site 0051), Lincoln, Rhode Island
  - Allergic Disease and Asthma Center ( Site 0027), Greenville, South Carolina
  - Diagnostics Research Group ( Site 0021), San Antonio, Texas
  - Allergy & Asthma Center ( Site 0001), Waco, Texas
  - Tidewater Physician Multispecialty Group, PC ( Site 0048), Williamsburg, Virginia
  - Bellingham Asthma & Allergy ( Site 0011), Bellingham, Washington
- Canada (3):
  - Recherche GCP Research ( Site 0802), Montreal, Quebec
  - Diex Recherche Quebec Inc ( Site 0805), Québec, Quebec
  - Clinique Specialisee en Allergie de la Capitale - CSAC ( Site 0800), Québec, Quebec
- Colombia (6):
  - Fundacion Centro de Investigacion Clinica CIC ( Site 0401), Medellín, Antioquia
  - Universidad Pontificia Bolivariana - Clinica Universitaria Bolivariana ( Site 0408), Medellín, Antioquia
  - MedPlus Medicina Prepagada S.A. ( Site 0402), Bogotá, Bogota D.C.
  - Centro Especializado en Enfermedades Pulmonares. ( Site 0410), Bogotá, Bogota D.C.
  - Healthy Medical Center S.A.S ( Site 0404), Zipaquirá, Cundinamarca
  - Instituto Neumologico del Oriente ( Site 0403), Floridablanca, Santander Department
- Germany (4):
  - Zentrum fuer ambulante pneumologische Forschung Marburg GbR ( Site 0910), Marburg, Hesse
  - Ballenberger Freytag Wenisch Institut fuer klinische Forschung GmbH ( Site 0917), Neu-Isenburg, Hesse
  - Pneumologicum im Suedstadtforum ( Site 0916), Hanover, Lower Saxony
  - Pneumologisches Studienzentrum ( Site 0911), Berlin
- Guatemala (6):
  - Celan SA ( Site 0500), Guatemala City
  - Clinica Medica Especializada en Neumologia y Tisiologia ( Site 0504), Guatemala City
  - Clinica Medica Especializada en Neumologia ( Site 0502), Guatemala City
  - Private Clinic ( Site 0505), Guatemala City
  - Clinica Privada Dr. Jose Francisco Flores Lopez ( Site 0503), Guatemala City
  - Instituto De Alergias y Enfermedades Respiratorias ( Site 0501), Guatemala City
- Peru (4):
  - Clinica Ricardo Palma ( Site 0601), San Isidro, Lima region
  - Asociacion Civil por la Salud ( Site 0602), Lima
  - Hospital Nacional Arzobispo Loayza ( Site 0607), Lima
  - Clinica Belen ( Site 0604), Piura
- Poland (9):
  - Centrum Medyczne Pratia Bydgoszcz ( Site 1206), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczny osrodek .All-Med. Grazyna Pulka ( Site 1203), Krakow, Lesser Poland Voivodeship
  - NZOZ CENTRUM ALERGOLOGII ( Site 1207), Lublin, Lublin Voivodeship
  - RCMed ( Site 1202), Sochaczew, Masovian Voivodeship
  - Centrum Medyczne Puławska ( Site 1215), Warsaw, Masovian Voivodeship
  - Centrum Medyczne Lucyna Andrzej Dymek - Zawadzkie ( Site 1200), Zawadzkie, Opole Voivodeship
  - Centrum Medyczne Pratia Katowice ( Site 1205), Katowice, Silesian Voivodeship
  - Centrum Medyczne Silmedic Sp z o o ( Site 1204), Katowice, Silesian Voivodeship
  - Gyncentrum Clinic Sp. z o.o. ( Site 1208), Katowice, Silesian Voivodeship
- Russia (16):
  - RSBHI Belgorod regional clinical hospital of Prelate Ioasafa ( Site 1417), Belgorod, Belgorod Oblast
  - GBUZ Regional Clinical Hospital 3 ( Site 1421), Chelyabinsk, Chelyabinsk Oblast
  - City Clinical Hospital No. 3 them. M. A. Podgorbunskogo ( Site 1401), Kemerovo, Kemerovo Oblast
  - Moscow City Clinical Hospital Number 13 ( Site 1460), Moscow, Moscow
  - Open Joint Stock Company Clinical and Diagnostic Center Euromedservice ( Site 1467), Moscow, Moscow
  - Clinic of FSBEI HE OmSMU of Minzdrav ( Site 1439), Omsk, Omsk Oblast
  - SPb SBHI City Consultative Diagnostic Center 1 ( Site 1409), Saint Petersburg, Sankt-Peterburg
  - GBUZ LO Center of Occupational Pathology ( Site 1447), Saint Petersburg, Sankt-Peterburg
  - Limited Liability Company Kurator ( Site 1425), Saint Petersburg, Sankt-Peterburg
  - SEIHPE Saint Petersburg SMU ( Site 1435), Saint Petersburg, Sankt-Peterburg
  - advisory diagnostic center No.85 ( Site 1455), Saint Petersburg, Sankt-Peterburg
  - Saratov City Clinical Hospital 2 n.a. V.I. Razumovsky ( Site 1453), Saratov, Saratov Oblast
  - Family Clinic ( Site 1465), Yekaterinburg, Sverdlovsk Oblast
  - State health Agency Ulyanovsk regional clinical hospital ( Site 1415), Ulyanovsk, Ulyanovsk Oblast
  - Voronezh Regional Clinical Hospital #1 ( Site 1441), Voronezh, Voronezskaja Oblast
  - SBCIH of the Yaroslavl region Central city hospital ( Site 1429), Yaroslavl, Yaroslavl Oblast
- South Korea (5):
  - Wonju Severance Christian Hospital ( Site 1502), Wŏnju, Kang-won-do
  - Asan Medical Center ( Site 1505), Songpagu, Seoul
  - Seoul National University Hospital ( Site 1501), Seoul
  - Severance Hospital Yonsei University Health System ( Site 1503), Seoul
  - Konkuk University Medical Center ( Site 1504), Seoul
- Spain (5):
  - Hospital Parc Tauli ( Site 1821), Sabadell, Barcelona
  - Hospital Clinico Universitario de Santiago ( Site 1820), Santiago de Compostela, La Coruna
  - Hospital General Universitario Gregorio Maranon ( Site 1823), Madrid, Madrid, Comunidad de
  - Hospital Ramon y Cajal ( Site 1815), Madrid
  - Hospital Clinico San Carlos ( Site 1822), Madrid
- Ukraine (14):
  - Kherson City Clinical Hospital n.a. Y.Y. Karabelesh ( Site 2811), Kherson, Kherson Oblast
  - F.G.Yanovskyy Institute of Phthisiology and Pulmonology ( Site 2802), Kyiv, Kyivska Oblast
  - F.G.Yanovskyy Institute of Phthisiology and Pulmonology ( Site 2808), Kyiv, Kyivska Oblast
  - SE Road Clinical Hospital 2 of Kyiv station ( Site 2812), Kyiv, Kyivska Oblast
  - SE O.S.Kolomiychenko Institute of Otolaryngology of NAMS of Ukraine ( Site 2817), Kyiv, Kyivska Oblast
  - Odesa regional clinical hospital ( Site 2804), Odesa, Odesa Oblast
  - City Polyclinic N20 ( Site 2806), Odesa, Odesa Oblast
  - Poltava City Clinical Hospital -1 ( Site 2813), Poltava, Poltava Oblast
  - Private Small-Scale Enterprise Medical Centre "Pulse" ( Site 2809), Vinnytsia, Vinnytsia Oblast
  - Vinnytsia Regional Clinical Hospital n.a. M.I. Pyrogov ( Site 2814), Vinnytsia, Vinnytsia Oblast
  - Volyn Regional Clinical Hospital ( Site 2816), Lutsk, Volyn Oblast
  - MI Zaporizhzhia City Multispecialty Clinical Hospital 9 ( Site 2803), Zaporizhzhia, Zaporizhzhia Oblast
  - Zhytomyr Central City Hospital No. 1 ( Site 2807), Zhytomyr, Zhytomyr Oblast
  - Medical Center of LLC Medical Clinic Blahomed ( Site 2815), Kyiv
- United Kingdom (4):
  - MeDiNova Yorkshire Dedicated Research Centre ( Site 2715), Shipley, Bradford
  - West Walk Surgery ( Site 2700), Yate, Gloucestershire
  - Medinova South London Research Centre ( Site 2706), Orpington, Kent
  - Medinova North London Dedicated Research Centre ( Site 2705), Northwood

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] McGarvey L, Sher M, Shvarts YG, Lu S, Wu WC, Xu P, Schelfhout J, La Rosa C, Nguyen AM, Reyfman PA, Afzal AS. The Efficacy and Safety of Gefapixant in a Phase 3b Trial of Patients with Recent-Onset Chronic Cough. Lung. 2023 Apr;201(2):111-118. doi: 10.1007/s00408-023-00606-w. Epub 2023 Mar 6. PMID 36879087

RESULTS

PARTICIPANT FLOW:
Groups:
- Gefapixant: Participants receive gefapixant at a dose of 45 mg administered as an oral tablet twice daily for 12 weeks.
- Placebo: Participants receive placebo matching gefapixant, administered as an oral tablet twice daily for 12 weeks.
Period: Overall Study
Arm/Group | Gefapixant | Placebo
Started | 208 | 211
Treated | 206 | 209
Completed | 192 | 201
Not Completed | 16 | 10
Not completed — Adverse Event | 2 | 1
Not completed — Death | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gefapixant | Placebo | Total
Number analyzed (Participants) | 208 | 211 | 419
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.6 (13.8) | 52.5 (13.7) | 52.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 135 | 271
  Male | 72 | 76 | 148
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 71 | 76 | 147
  Not Hispanic or Latino | 136 | 134 | 270
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 22 | 28 | 50
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 151 | 152 | 303
  More than one race | 29 | 29 | 58
  Unknown or Not Reported | 0 | 0 | 0
Baseline Leicester Cough Questionnaire (LCQ) [Mean (Standard Deviation); unit: Scores on a scale] — The LCQ is a 19-item, cough-specific health related qualify of life (HRQoL) questionnaire. Each item on the LCQ assesses symptoms using a 7-point scale ranging from 1 to 7. The LCQ contains three domains on physical, psychological, and social functioning, and each domain score is calculated as the mean score of the items (range: 1 to 7) within the domain. The LCQ total score is the sum of the 3 domains, with a range from 3 (lowest total score) to 21 (highest total score). Higher scores indicate better HRQoL Population: Includes randomized participants who had LCQ total score values at baseline
  Scores on a scale
    number analyzed (Participants) | 202 | 200 | 402
    (all) | 10.8 (3.1) | 11.3 (2.8) | 11.0 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Leicester Cough Questionnaire (LCQ) Total Score at Week 12
Description: Participants will be asked to complete the LCQ to assess the impact of their cough severity on health related quality of life (HRQoL) over the past 2 weeks. The LCQ is a 19-item, cough-specific HRQoL questionnaire. Each item on the LCQ assesses symptoms using a 7-point scale ranging from 1 to 7. The LCQ contains three domains on physical, psychological, and social functioning, and each domain score is calculated as the mean score of the items (range: 1 to 7) within the domain. The LCQ total score is the sum of the 3 domains, with a range from 3 (lowest total score) to 21 (highest total score). Higher scores indicate better HRQoL. The change from baseline in LCQ total score is calculated.
Time Frame: Baseline, Week 12
Population: All randomized participants who have taken at least one dose of study intervention, and had LCQ total score values at both baseline and week 12. Participants were analyzed in the group as randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 199 | 199
Scores on a Scale | 4.34 [3.84 to 4.83] | 3.59 [3.09 to 4.09]
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Superiority; p = 0.034, Longitudinal ANCOVA; The model included terms for treatment group, visit, interaction of treatment by visit, gender, and baseline LCQ total score; Estimated difference = 0.75, 95% CI 2-sided [0.06 to 1.44] — The estimated difference is the treatment difference in model based mean change from baseline at Week 12

2. Secondary Outcome: Change From Baseline in the Cough Severity Visual Analog Scale (VAS) Score at Week 12
Description: Participants will be asked to complete the VAS questionnaire to assess the severity of their cough over the past 24-hours. The Cough Severity VAS is a single-item questionnaire asking the participant to rate the severity of their cough on a 100-point scale ranging from 0 ("No Cough") to 100 ("Extremely Severe Cough"). Higher scores indicate greater severity of cough. The change from baseline in VAS score is calculated.
Time Frame: Baseline, Week 12
Population: All randomized participants who have taken at least one dose of study intervention, and had VAS total score values at both baseline and week 12. Participants were analyzed in the group as randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 201 | 205
Scores on a Scale | -31.79 [-35.37 to -28.20] | -24.87 [-28.41 to -21.32]
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Other; p = 0.006, Longitudinal ANCOVA — Nominal p value, not controlled for multiplicity; The model included terms for treatment group, visit, interaction of treatment by visit, gender, and baseline mean weekly cough severity VAS score; Estimated Difference = -6.92, 95% CI 2-sided [-11.88 to -1.97] — The estimated difference is the treatment difference in model based mean change from baseline at Week 12

3. Secondary Outcome: Percentage of Participants With One or More Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants with one or more AEs is presented.
Time Frame: Up to approximately 14 weeks
Population: All randomized participants who received at least 1 dose of study intervention. Participants were analyzed in the group as treated.
Measure: Number; unit: Percentage of Participants
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 206 | 209
Percentage of Participants | 65.5 | 43.1

4. Secondary Outcome: Percentage of Participants Who Discontinue Study Drug Due to an AE
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinue study drug due to an AE is presented.
Time Frame: Up to approximately 12 weeks
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 206 | 209
Percentage of Participants | 11.2 | 1.9

ADVERSE EVENTS:
Time Frame: Up to 114 days
Description: All-cause mortality population includes all randomized participants. Serious and other adverse events population includes all participants who received at least 1 dose of study intervention. Participants were analyzed in the group as treated.
Arm/Group | Gefapixant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/208 | 1/211
Serious Adverse Events (participants affected / at risk) | 3/206 | 4/209
Other Adverse Events (participants affected / at risk) | 105/206 | 22/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefapixant (N=206) | Placebo (N=209)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Tonsillar cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefapixant (N=206) | Placebo (N=209)
Ageusia (Nervous system disorders) | 24 (24) | 0 (0)
Dysgeusia (Nervous system disorders) | 66 (70) | 7 (7)
Headache (Nervous system disorders) | 11 (12) | 14 (15)
Hypogeusia (Nervous system disorders) | 22 (22) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT04193202/Prot_SAP_000.pdf